CLINICAL TRIAL: NCT01017510
Title: Comparative Study Examining the Effectiveness in Use of a DERMOJET and a Normal Syringe Treatment for Patients With Hair Loss - Alopecia Areata
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Dr. Boaz Ami-Chi, Dermatology Dept Sheba Medical Center
Model: Parallel | Masking: None
Other Study IDs: SHEBA-09-7322-BA-CTIL
Record Dates: First submitted 2009-11-18; First posted 2009-11-20 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Subcutaneous injection luer syringe — Right scalp: Luer syringe.
  Left scalp: syringe without a needle.
  All injections will contain 0.1 ml of Depo Medrol - Methylprednisolone acetate 40 mg/2 ml.
  The distance between injection locations will be 1 cm.
Device: DERMOJET (a syringe without a needle) — Right scalp: Luer syringe.
  Left scalp: syringe without a needle.
  All injections will contain 0.1 ml of Depo Medrol - Methylprednisolone acetate 40 mg/2 ml.
  The distance between injection locations will be 1 cm.

SUMMARY:
Conventional treatments include the use of steroids applied locally, or injection in to the legion, or oral therapy.

Treatment is determined by the severity of the disease.

Injection in to the legion can be done in two methods

1. Subcutaneous injection syringe Lower
2. Using syringe DERMOJET - a syringe without a needle. So far there are no publications in the medical literature of studies comparing efficacy, safety, convenience of use for doctor-patient, of both methods.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects over the age of 18
2. Men and women
3. The presence of at least two lesions (centers) in diameter of at least 1.5 cm on both sides of the scalp.
4. Healthy with no diseases that constitute the background against the total label use steroids

Exclusion Criteria:

1. Pregnant women
2. Involvement of more then 50% of the scalp
3. Patients with immunodeficiency-related diseases
4. Patients receiving systemic steroids

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2009-11; Primary Completion 2010-11 (Estimated); Study Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Evaluation of lesions will be based on Global assessment of improvement, score of 0-5 | 1 year

SECONDARY OUTCOMES:
Pain level will be evaluated based on a scale of 0-10 | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: BOAZ AMI-CHI, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Rmat Gan, Israel